CLINICAL TRIAL: NCT06710002
Title: Effectiveness of a Telerehabilitation Program for Improving Sexual Function and Reducing Pain in Menopausal Women With Dyspareunia: Protocol of a Randomized Clinical Trial.
Brief Title: Effectiveness of a Telerehabilitation Program for Improving Sexual Function and Reducing Pain in Menopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Médico Tecnológico SL (Other)
Collaborators: RAPbarcelona (Other)
Responsible Party: Principal Investigator, Inés Ramírez García, Principal Investigator. Professor. Physiotherapist PhD, University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAPbarcelonaPAULA
Record Dates: First submitted 2024-11-18; First posted 2024-11-29 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Menopause; Genitourinary Syndrome of Menopause; Dyspareunia
Keywords: Physiotherapy; Telerehabilitation; face to face treatment; female sexual function; vaginal dilators; manual therapy; capacitive resistive monopolar radiofrequency
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Asynchronous Online Telerehabilitation Program (Experimental): For this study, a five weeks course called "Pelvify: Menopause and dyspareunia treatment" will be created. This will be based on a set of explanatory and demonstrative videos focused on self-treatment of pain during sexual intercourse.
  Each patient will have an individual access (own user). All groups in the sixth week will have a face-to-face visit to assess their progress. A telephone follow-up will be carried out at six months and twelve months after the end of the treatment.
  Interventions: Behavioral: Pelvify: Menopause and dyspareunia treatment
- Face to Face Physical Therapy Protocol (Active Comparator): This consists of carrying out 5 individual sessions of 45 minutes, 1 day a week at the physiotherapy clinic RAPbarcelona S.L.
  Patients will be placed comfortably supine with a pillow under their head, with their legs flexed on two leg warmers, in the lithotomy position, without underwear and covered with a drape.
  In each of the treatment sessions, the same structure will always be applied and the established protocol will be followed.
  All groups in the sixth week will have a face-to-face visit to assess their progress. A telephone follow-up will be carried out at six months and twelve months after the end of the treatment.
  Interventions: Other: Face to Face Physical Therapy Protocol
- Face to Face Protocol Combined With an Asynchronous Telerehabilitation Program (Active Comparator): This group will carry out the same 5 individual sessions of 45 minutes, 1 day a week at the RAPbarcelona S.L physiotherapy clinic following the protocol described for the "Face to Face Physical Therapy Protocol" group and in addition to the first visit they will be given access and instructions to follow in parallel the asynchronous online telerehabilitation program "Pelvify: Menopause and dyspareunia treatment".
  All groups in the sixth week will have a face-to-face visit to assess their progress. A telephone follow-up will be carried out at six months and twelve months after the end of the treatment.
  Interventions: Other: Face to Face Protocol Combined With an Asynchronous Telerehabilitation Program

INTERVENTIONS:
Behavioral: Pelvify: Menopause and dyspareunia treatment — Topics addressed in the Asynchronous Online Telerehabilitation Program would be:
  1. What it is and why it hurts during sex. What is dyspareunia?
  2. How to recover vaginal elasticity.
  3. Massage
  4. Self-palpation.
  5. Stretching of the pelvic floor muscles.
  6. Use of vaginal dilators.
  7. Moisturizers and lubricants.
  8. Sexual pleasure.
  9. Communication with the partner.
  Arms: Asynchronous Online Telerehabilitation Program
Other: Face to Face Physical Therapy Protocol — Physical Therapy Protocol will be based on:
  1. Health education:
  2. CMRF: INDIBA® ACTIV CT8 will be used to apply the radiofrequency
  3. Manual therapy: it will be based on performing the Thiele's massage.
  4. Vaginal dilators: FEMINAFORM® vaginal dilators will be used.
  Arms: Face to Face Physical Therapy Protocol
Other: Face to Face Protocol Combined With an Asynchronous Telerehabilitation Program — Both, the face to face protocol and the Asynchronous Telerehabilitation Program will be carried on on this group.
  Arms: Face to Face Protocol Combined With an Asynchronous Telerehabilitation Program

SUMMARY:
The aim of this study is to analyze the effectiveness of a telerehabilitation program with respect to a face-to-face physiotherapy protocol in relation to the improvement of sexual function, the reduction of pain and the improvement of the quality of life, in the treatment of menopausal women with dyspareunia.

DETAILED DESCRIPTION:
Both therapies have been proven to be effective, but since now any randomized controlled trial has been conducted to compare the results regarding the improvement in the sexual function, the reduction of pain and the improvement of quality of life in this population. The investigators hypothesize that the implementation of an asynchronous online telerehabilitation program is not inferior to the effect of the treatment carried out with a face-to-face physiotherapy protocol, in relation to the main variables obtained with the instruments Female Sexual Function Index (FSFI), the Visual Analogue Scale (VAS) and Menopause Specific Quality of Life Questionnaire (MENQOL). Secondary goals are: 1) to evaluate whether the incorporation of a telerehabilitation program to face-to-face treatment increases the effectiveness in relation to performing only the face-to-face physiotherapy protocol, 2) compare the size of the vaginal dilator inserted painlessly at the end of the treatment in all groups, 3) identify any adverse effects associated with the intervention during the study, 4) detail the degree of adherence to the treatment and 5) record satisfaction with the treatment using the Likert Scale.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age from 45 to 65 years.
* Menopausal
* Suffer dyspareunia for 3 months of evolution.
* Willing to complete study questionnaires and informed consent study.

Exclusion Criteria:

* Pacemaker or other types of electronic implant.
* Thrombophlebitis.
* Skin hypersensitivity or rejection of manual contact.
* Active or previous treatment with chemotherapy or radiotherapy in the pelvic area.
* Wounds or burns in the pelvic area.
* Allergy to nickel and chromium.
* Other pelvic floor physiotherapy treatments during the study intervention.
* Other medical and surgical treatments in the pelvic region, such as muscle infiltrations or nerve blocks during the study intervention.
* Surgical intervention in the pelvic area in the last 3 months.
* Fibromyalgia.
* Oncological processes that affect the sacrum.
* Systemic diseases (infectious, vascular, endocrine, metabolic or neoplastic conditions).
* Neuromuscular diseases (Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Myasthenia Gravis or spinal muscular atrophy).
* Myelopathy and Osteomyelitis.
* Diseases that cause alterations of the central nervous system (traumatic or vascular spinal cord injury).
* Neurological or metabolic conditions that affect the ability to respond (Diabetes, Parkinson's disease, senile dementia, etc).
* Serious mental disorder.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Improved Female Sexual Function via Female Sexual Function Index (FSFI) | From registration to the end of treatment at 5 weeks, one week after the end of treatment, and at 6 and 12 months post-treatment
  FSFI it is a self-administered instrument made up of 19 questions grouped into 6 domains: desire, arousal, lubrication, orgasm, satisfaction and pain. Response is measured on a scale from 0 (no sexual activity) to 5 (almost always). The FSFI total score range is 2 to 36; a score of less than or equal to 26.55 points, or when the score of any domain is less than 3.6 points, is considered a risk criterion for sexual dysfunction.
Reduction in the Intensity of Dyspareunia Pain via Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 5 weeks, one week after treatment, and at six months and twelve months post treatment
  This scale (VAS) adequately captures the intensity of pain perceived by the patient represented by a horizontal line of 10 cm, where the left end (0 cm) is the absence of pain and the right end (10 cm) is pain of maximum intensity possible. The patient is asked to mark on the line the point indicating the intensity of their pain and it is measured with a millimeter ruler. The intensity is expressed in centimeters. It is considered mild up to 4 cm, moderate from 5 to 7 cm and if it is greater than 7 cm.
Improved Quality of Life via Menopause Specific Quality of Life Questionnaire (MENQOL) | From registration to the end of treatment at 5 weeks, one week after the end of treatment, and at 6 and 12 months post-treatment
  MENQOL it is a questionnaire designed to assess the quality of life of women who are going through menopause. It consists of 29 questions grouped into 4 domains: vasomotor area, psychosocial area, physical area and sexual area. Each question has two answer options No/Yes, if yes, it is assigned a score ranging from 0 (not annoying) to 6 (very annoying). The total score is from 29 to 232 points. A higher score indicates more intense symptomatology.

SECONDARY OUTCOMES:
Change from the size of the Vaginal Dilator inserted without pain | From enrollment to one week after treatment
  It will be measured with FEMINAFORM® vaginal dilators. The set consists of 4 dilators of different diameters and lengths, and a clamping device: Size 1: 22mmx85mm (diameter/length), Size 2: 27x105mm (diameter/length), Size 3: 32x135mm (diameter/length) and Size 4 : 37x160mm (diameter/length).
  The largest vaginal dilator size that has a score (VAS) of 0 cm will be recorded. It will be specified whether the absence of pain is by inserting the entire dilator or only a part.

OTHER OUTCOMES:
Number of complaints or adverse effects registered during treatments | During the five weeks of treatment and one week after finishing it.
  Any type of discomfort or alteration of normality during the application or after the end of the treatment, will be recorded
Degree of Satisfaction Score on the treatment using the Likert Scale. | One week after the end of treatment, and 6 months and 12 months after treatment
  The six-point Likert Scale is a psychometric measurement tool that assesses subjective attitudes and opinions. Each level of the scale is given a numerical value. It will be expressed as: 1 = Strongly Disagree, 2 = Disagree, 3 = Slightly Disagree, 4 = Slightly Agree, 5 = Agree and 6 = Strongly Agree.
Degree of Adherence to the treatments | During the five weeks of treatment, 1 week after treatment, and at 6 months and 12 months after treatment
  Monitored by tracking attendance at treatment sessions according to the following scale: 1 = No adherence (less than 20%), 2 = Minimal adherence (20% - 39%), 3 = Low adherence (40% - 59%), 4 = Moderate adherence (60% - 79%), 5 = High adherence (80% - 99%), and 6 = Complete adherence (100%).

CONTACTS AND LOCATIONS:
Locations (1):
- RAPbarcelona, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marino JM. Genitourinary Syndrome of Menopause. J Midwifery Womens Health. 2021 Nov;66(6):729-739. doi: 10.1111/jmwh.13277. Epub 2021 Aug 31. PMID 34464022